CLINICAL TRIAL: NCT06030648
Title: Intravenous Administration of Mesenchymal Stem Cells (IV-MSC) for the Treatment of Cerebral Adrenoleukodystrophy (cALD)
Brief Title: MT2022-01: MSCs for ALD
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Awaiting supplies
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022LS001
Record Dates: First submitted 2023-08-31; First posted 2023-09-11 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cerebral Adrenoleukodystrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV-MSC for cALD (Early Disease/Bridge Therapy) (Experimental): Patients with active, cerebral adrenoleukodystrophy (cALD) as a bridge to hematopoietic stem cell transplant or gene therapy.
  Interventions: Biological: Mesenchymal stem cells (IV-MSC)
- IV-MSC for cALD (Advanced Disease) (Experimental): Patients with active, cerebral adrenoleukodystrophy (cALD) who are too advanced for gene therapy or HSCT.
  Interventions: Biological: Mesenchymal stem cells (IV-MSC)

INTERVENTIONS:
Biological: Mesenchymal stem cells (IV-MSC) — Patients will receive 1 infusion (1 x 106 cells/kg on day 0) then be followed for 8 weeks from the infusion.

SUMMARY:
This is a single-institution study to evaluate the use of intravenously administered allogeneic, 3rd party mesenchymal stem cells (IV-MSC) in patients with active, cerebral adrenoleukodystrophy (CALD), as a bridge to hematopoietic stem cell transplant or gene therapy, or in patients who are too advanced for gene therapy or HSCT. The intervention will occur in the time between diagnosis of active CALD and transplant which is currently 8-12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 3 years
* diagnosis of ALD, as established by elevation of very long chain fatty acid levels or gene mutation
* evidence of active cerebral disease as determined by the presence of gadolinium enhancement
* ALD MRI (Loes) score ≥ 1
* Patients who have not received prior gene therapy or transplant
* Life expectancy of > 6 months as determined by the enrolling researcher
* Have adequate organ function confirmed by laboratory values obtained within 28 days prior to enrollment

Exclusion Criteria:

* Inability to undergo sedation or MRI studies for any reason
* Other concurrent life-threatening disease (life expectancy <6 months) or eligible for hospice care
* Known or suspected hypersensitivity to human serum albumin, diphenhydramine, acetaminophen, methylprednisolone, or any of the components of IMS001.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of intravenously-administered allogeneic, third-party mesenchymal stem cells (IV-MSC). | 6 months
  Safety and tolerability of cerebral adrenoleukodystrophy (cALD) patients receiving intravenously-administered allogeneic, third-party mesenchymal stem cells (IV-MSC) assessed by incidence of adverse events.

SECONDARY OUTCOMES:
Incidence of radiographic response in patients receiving intravenously-administered allogeneic, third-party mesenchymal stem cells (IV-MSC). | 6 months
  Radiographic response is defined as the resolution of intravenous gadolinium contrast enhancement on brain MRI.

CONTACTS AND LOCATIONS:
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States